CLINICAL TRIAL: NCT03933618
Title: A Randomized Double Blinded Placebo Controlled Trial Between Anastrozole and Clomiphene to Evaluate Improvement in Hypogonadal Symptoms and Erectile Function Using ADAM, IIEF and EHS Validated Scales
Brief Title: Anastrazole and Clomiphene to Evaluate Hypogonadal Symptoms and Erectile Function
Acronym: CAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 4134
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Anastrozole; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (6):
- anastrazole-clomiphene-placebo (Other): anastrozole for eight weeks then clomiphene for eight weeks then placebo for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap
- anastrazole-placebo-clomiphene (Other): anastrozole for eight weeks then placebo for eight weeks then clomiphene for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap
- clomiphene-anastrazole-placebo (Other): clomiphene for eight weeks then anastrozole for eight weeks then placebo for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap
- clomiphene-placebo-anastrazole (Other): clomiphene for eight weeks then placebo for eight weeks then anastrozole for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap
- placebo-clomiphene-anastrazole (Other): placebo for eight weeks then clomiphene for eight weeks then anastrozole for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap
- placebo-anastrazole-clomiphene (Other): placebo for eight weeks then anastrozole for eight weeks then clomiphene for eight weeks
  Interventions: Drug: Anastrozole 1mg; Drug: Clomiphene Citrate 25mg; Drug: Placebo - Cap

INTERVENTIONS:
Drug: Anastrozole 1mg
Drug: Clomiphene Citrate 25mg
Drug: Placebo - Cap

SUMMARY:
This study evaluates anastrazole and clomiphene in the improvement in hypogonadal symptoms and erectile function. Each subject will receive Anastrazole 1 mg/day, clomiphene 25 mg/day and placebo in randomized schedule of 8 week intervals.

DETAILED DESCRIPTION:
Aromatase inhibitors (AI) (Anastrazole) and selective estrogen receptor modifiers (SERMS)(clomiphene) increase testosterone production through stimulation of the hypothalamic pituitary axis. While these drugs both reduce the feedback inhibition of estrogen on the pituitary, SERMs cause an increase in serum estradiol, whereas AIs reduce estradiol levels. Using these medications, we can obtain therapeutic testosterone levels with either an increase or decrease in estradiol levels.

ELIGIBILITY:
Inclusion Criteria:

1. Men age 18-70
2. Baseline morning Testosterone 150-350 ng/dL x2
3. leutenizing hormone (LH) 1.5-9.2 miU/mL, Follicle stimulation hormone (FSH) 1.6-8.0 miU/mL, Prolactin 4-15 ng/mL
4. Positive Androgen Deficiency in the Aging Male (ADAM) score. A positive score is when an affirmative answer (''yes'') to either questions "Do you have a decreased sex drive/libido?" or "Are your erections less strong?" or any three other questions.10
5. Body mass index (BMI) <40
6. Sexual health inventory for men (SHIM) score >7 and <21. Patients are allowed to be taking phosphodiesterase 5 inhibitors (i.e. Viagra, Levitra, Cialis) at baseline, however we will ask them to do the SHIM survey as if they were not taking this medication.
7. Men must attempt to have at least four sexual encounters over each of the eight-week periods
8. Men willing not to take phosphodiesterase 5 inhibitors throughout the entire study

Exclusion Criteria:

1. Current or previous history of prostate cancer
2. Previous or current androgen deprivation therapy for prostate cancer,
3. Past surgical history of prostatectomy.
4. History of testicular cancer.
5. History of deep vein thrombosis (DVT) or blood dyscrasia
6. History of breast cancer
7. Men with past or current treatment for erectile dysfunction including MUSE (alprostodil), intracavernosal injections, penile prosthesis. Men not on treatment or men who are on phosphodiesterase inhibitors will be allowed to be in the study but must stop their use at the screening visit.
8. Chronic opioid use
9. Use of steroids within the past 3 months, including prednisone and/or cortisone injections, and inhaled steroids. Topical steroid cream is acceptable.
10. History of or current use of anabolic steroids, i.e. testosterone, (or any analog of testosterone) dihydroepiandrosterone (DHEA), dihydroepiandrosterone sulfate (DHEAS) or any growth promoters i.e. growth hormone itself or analogs of growth hormone
11. History of or current use of anti-androgen medications, i.e. Aldactone, Tagamet, estrogens
12. Alcohol intake > 30 grams (drink more than 2 beers per day OR more than 1 glass of wine or cocktail daily)
13. Having started a new medication during the past three months which may interfere with the outcome measures of the study
14. Polycythemia (HCT >52% )
15. History of prostate specific antigen (PSA)> 4.0 ng/dl
16. Hematocrit (HCT)< 36 %
17. Liver function tests greater than 2 times upper normal limits or history of abnormal electrolytes, calcium or Parathyroid hormone without workup, at the discretion of the investigator.
18. Previous hypogonadal treatment within last 3 months. -

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Welliver, MD, Principal Investigator — Albany Medical College

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men will be incentivized to come to each clinic appointment with $20 dollars at the end. If they complete the study they will be able to earn $100. Men will be incentivized to not use phosphodiesterase inhibitors throughout the study by giving them three 100mg tablets of Viagra per month of the study for a total of twelve 100 mg tablets.
Groups:
- Anastrazole-clomiphene-placebo: anastrozole for eight weeks then clomiphene for eight weeks then placebo for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
- Anastrazole-placebo-clomiphene: anastrozole for eight weeks then placebo for eight weeks then clomiphene for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
- Clomiphene-anastrazole-placebo: clomiphene for eight weeks then anastrozole for eight weeks then placebo for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
- Clomiphene-placebo-anastrazole: clomiphene for eight weeks then placebo for eight weeks then anastrozole for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
- Placebo-clomiphene-anastrazole: placebo for eight weeks then clomiphene for eight weeks then anastrozole for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
- Placebo-anastrazole-clomiphene: placebo for eight weeks then anastrozole for eight weeks then clomiphene for eight weeks
  Anastrozole 1mg
  Clomiphene Citrate 25mg
  Placebo - Cap
Period: Baseline
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Baseline to Week 8
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 8 to Week 16
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 16 to Week 24
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 4 | 4 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 4 | 3 | 4 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: IIEF (International Index of Erectile Function) Score - Screen
Description: 15 item self reported erectile function. Each item is scored 0-5 with 0=negative response and 5 = positive response with totals of 0-75
Time Frame: At baseline
Population: Total IIEF reported at the initial encounter.
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 34 | 43 | 57 | 41 | 57 | 24
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 57 | 57 | 45 | 32 | 36 | 55
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 55 | 46 | 41 | 45 | 58 | 32
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 | 50 | 52 | 55 | 47 | 18 | 62

2. Primary Outcome: IIEF (International Index of Erectile Function) Score - Week 8
Description: 15 item self reported erectile function over the past 8 weeks. Each item is scored 0-5 with 0=negative response and 5 = positive response with totals of 0-75
Time Frame: Week 8
Population: Total IIEF reported at the end of the first 8 week period
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 25 | 55 | 32 | 20 | 66 | 35
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 45 | 51 | 63 | 45 | 72 | 37
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 55 | 59 | 32 | 65 | 43 | 28
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 | 63 | 65 | 70 | 45 | 25 | 53

3. Primary Outcome: IIEF (International Index of Erectile Function) Score - Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Total IIEF reported at the end of the second 8 week period - at week 16
  Data for patient 23 was not collected in the placebo-clomiphene-anastrazole arm.
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 45 | 53 | 35 | 45 | 66 | 37
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 43 | 56 | 50 | 55 | 33 | 38
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 53 | 62 | 37 | 58 | 59 | 15
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 62 | 38 | 51 | 47 |  | 18

4. Primary Outcome: IIEF (International Index of Erectile Function) Score - Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: Total IIEF reported at the end of the final 8 week period - at week 24
  Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 12 | 70 | 42 | 52 | 65 | 41
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 54 | 60 | 43 | 35 | 27 | 45
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 60 | 65 |  | 72 | 45 | 17
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 52 | 59 | 60 | 47 |  | 14

5. Secondary Outcome: Normalized Testosterone - Screen
Description: Normalized at >350ng/dl
Time Frame: Baseline
Population: Normalized Testosterone measured week 0 - initial screen
  Data not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 205 | 330 | 226 | 367 | 315 | 321
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 293 | 237 | 194 | 300 | 214 | 243
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 347 | 328 | 268 | 206 | 321 | 148
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 95 | 291 | 306 | 244 |  | 289

6. Secondary Outcome: Normalized Testosterone - Week 8
Description: Normalized at >350ng/dl
Time Frame: Week 8
Population: Normalized Testosterone measured at the end of the first 8 week period
  Data for patient 23 was not collected for placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 484 | 757 | 566 | 1316 | 133 | 470
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 387 | 296 | 693 | 917 | 271 | 298
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 607 | 453 | 216 | 527 | 270 | 139
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 545 | 676 | 592 | 497 |  | 296

7. Secondary Outcome: Normalized Testosterone - Week 16
Description: Normalized at >350ng/dl
Time Frame: Week 16
Population: Normalized Testosterone measured at the end of the 16th week
  Data for patient 23 was not collected for placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 437 | 591 | 338 | 391 | 696 | 502
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 337 | 200 | 451 | 403 | 396 | 520
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 329 | 191 | 124 | 206 | 585 | 283
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 609 | 323 | 456 | 288 |  | 484

8. Secondary Outcome: Normalized Testosterone - Week 24
Description: Normalized at >350ng/dl
Time Frame: Week 24
Population: Normalized Testosterone measured at the end of the 24th week
  Data was not collected for patient 15 clomiphene-anastrazole-placebo Data for patient 23 was not collected for placebo-clomiphene-anastrazole arm Data was not collected for patient 24 in placebo-anastrazole-clomiphene
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 268 | 793 | 214 | 537 | 412 | 596
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 269 | 519 | 440 | 531 | 375 | 972
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 446 | 449 |  | 447 | 487 | 195
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 196 | 630 | 274 | 486 |  |

9. Secondary Outcome: ADAM (Androgen Deficiency in the Aging Male) Score - Screen
Description: Self reported quantification of hypogonadism. 10 "yes" or "no" questions.
  A positive (yes) questionnaire result is defined as a "yes or 1" and a negative (no) questionnaire result is defined as a "no or 0" to question 1 or question 7 or any 3 other questions.
  Yes (1) represents a better outcome than No (1)
  In Data Entry:
  Yes - 1 No - 0
Time Frame: Baseline
Population: Initial Evaluation for ADAM score - Week 0
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 | 1 | 1 | 1 | 1 | 1 | 1

10. Secondary Outcome: ADAM (Androgen Deficiency in the Aging Male) Score - Week 8
Description: as for outcome 9
Time Frame: Week 8
Population: ADAM score at the end of Week 8
  Data was not collected for patient 19 in anastrazole-clomiphene-placebo arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 1 | 1 | 0 | 1 | 0 | 1
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1 | 0 | 1 | 0 | 0 | 1
  Patients 19-24: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 |  | 1 | 1 | 1 | 1 | 1

11. Secondary Outcome: ADAM (Androgen Deficiency in the Aging Male) Score - Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: ADAM score at the end of Week 16 Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 1 | 1 | 1 | 1 | 0 | 1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1 | 1 | 1 | 0 | 0 | 1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 1 | 1 | 1 | 1 |  | 1

12. Secondary Outcome: ADAM (Androgen Deficiency in the Aging Male) Score - Week 24
Description: as for outcome 9
Time Frame: Week 24
Population: ADAM score at the end of Week 24 No data collected pt 15 in clomiphene-anastrazole-placebo arm no data collected for pt 16 clomiphene-placebo-anastrazole arm no data collected for pt 23 placebo-clomiphene-anastrazole arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 1 | 0 | 0 | 1 | 0 | 1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 1
  Patients 13-18 | 0 | 0 |  |  | 1 | 1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 1 | 1 | 1 | 0 |  | 1

13. Secondary Outcome: EHS (Erectile Hardness Score) - Screen
Description: Self reported questionnaire rated 0-4 0=penis does not enlarge, 4=Penis completely hard and fully rigid
Time Frame: Baseline
Population: Score 0-4 at the initial encounter week 0
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3 | 3 | 3 | 2 | 3 | 3
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 3 | 3 | 3 | 2 | 3 | 3
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 3 | 3 | 3 | 2 | 1 | 3
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 | 3 | 3 | 3 | 3 | 3 | 3

14. Secondary Outcome: EHS (Erectile Hardness Score) - Week 8
Description: Self reported questionnaire rated 0-4 0=penis does not enlarge, 4=Penis completely hard and fully rigid
Time Frame: Week 8
Population: Score 0-4 at the end of Week 8
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 1 | 4 | 1 | 1 | 3 | 1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 3 | 3 | 3 | 2 | 4 | 2
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 3 | 3 | 3 | 3 | 1 | 3
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 19-24 | 3 | 3 | 3 | 2 | 1 | 3

15. Secondary Outcome: EHS (Erectile Hardness Score) - Week 16
Description: Self reported questionnaire rated 0-4 0=penis does not enlarge, 4=Penis completely hard and fully rigid
Time Frame: Week 16
Population: Score 0-4 at the end of Week 16
  Data for patient 23 was not collected in placebo-clomiphene-anastrazole arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3 | 3 | 2 | 2 | 4 | 3
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 3 | 3 | 3 | 3 | 2 | 3
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 3 | 4 | 3 | 4 | 1 | 0
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 3 | 1 | 3 | 3 |  | 1

16. Secondary Outcome: EHS (Erectile Hardness Score) - Week 24
Description: Self reported questionnaire rated 0-4 0=penis does not enlarge, 4=Penis completely hard and fully rigid
Time Frame: Week 24
Population: Score 0-4 at the end of Week 24 no data was collected for patient 15 in clomiphene-anastrazole-placebo no data was collected for patient 23 in placebo-clomiphene-anastrazole
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3 | 4 | 2 | 2 | 3 | 3
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 3 | 3 | 3 | 2 | 2 | 3
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 3 | 4 |  | 4 | 1 | 1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 3 | 1 | 3 | 3 |  | 1

17. Secondary Outcome: LH - Screen
Description: Luteinizing Hormone levels collected at the initial encounter and at the end of the 8, 16, and 24 week periods.
Time Frame: Baseline
Population: LH measured at initial encounter
  Data for pt 23 in placebo-clomiphene-anastrazole not collected
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3.5 | 3.6 | 3.8 | 6.8 | 3.5 | 3.4
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 3.4 | 3.8 | 2.4 | 4.1 | 2.4 | 1.7
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1.1 | 3.5 | 4.1 | 3.3 | 6 | 3.1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 6.3 | 4.1 | 4.7 | 5.9 |  | 6.8

18. Secondary Outcome: LH - Week 8
Description: Luteinizing Hormone levels collected at the initial encounter and at the end of the 8, 16, and 24 week periods.
Time Frame: Week 8
Population: LH measured at week 8
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 9.1 | 5.1 | 9.9 | 17.3 | 3.6 | 6.3
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 5.2 | 4 | 10.7 | 12.6 | 3.3 | 1.9
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 2.9 | 6.9 | 6.1 | 4.7 | 6.7 | 3
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 4.2 | 11.5 | 7.5 | 6.9 |  | 7.3

19. Secondary Outcome: LH - Week 16
Description: Luteinizing Hormone levels collected at the initial encounter and at the end of the 8, 16, and 24 week periods.
Time Frame: Week 16
Population: LH measured at week 16
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 6.8 | 4.6 | 4.2 | 5.4 | 13.9 | 8.9
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 6.9 | 4.8 | 6.3 | 4.9 | 5.2 | 3.8
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1.9 | 2.1 | 2.2 | 1.9 | 13 | 6.4
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 7.8 | 4.3 | 6.6 | 4.9 |  | 7.4

20. Secondary Outcome: LH - Week 24
Description: Luteinizing Hormone levels collected at the initial encounter and at the end of the 8, 16, and 24 week periods.
Time Frame: Week 24
Population: LH measured at week 24
  No data for patient 13 collected in clomiphene-anastrazole-placebo arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm Data was not collected for patient 24 in placebo-anastrazole-clomiphene arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3 | 4.1 | 3.4 | 6.4 | 5 | 7.7
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 6.1 | 12.6 | 5.9 | 6.4 | 2.9 | 10.5
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 2.2 | 5.4 |  | 7.6 | 7.1 | 8.1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 2.7 | 15.1 | 4.7 | 5.4 |  |

21. Secondary Outcome: FSH - Screen
Description: Lab Values for follicle stimulating hormone
Time Frame: Baseline
Population: FSH measured at initial encounter
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 2.7 | 2.4 | 5.5 | 4.5 | 3.3 | 3.6
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 5.7 | 3.7 | 3.9 | 2.9 | 1.8 | 3.5
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1.6 | 5.1 | 1.7 | 4 | 4.4 | 5.7
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 5.5 | 10 | 4.5 | 4.4 |  | 5.1

22. Secondary Outcome: FSH - Week 8
Description: Lab Values for follicle stimulating hormone
Time Frame: Week 8
Population: FSH measured at Week 8
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 5.4 | 4.3 | 8.2 | 16.2 | 3.4 | 4.1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 7.7 | 6.2 | 7.8 | 3.03 | 2.2 | 4.2
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 3 | 8.3 | 1.8 | 6.3 | 4.7 | 6
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 11.3 | 20.3 | 6.1 | 8.1 |  | 4.4

23. Secondary Outcome: FSH - Week 16
Description: Lab Values for follicle stimulating hormone
Time Frame: Week 16
Population: FSH measured at Week 16
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 7 | 4.3 | 4.2 | 5.3 | 10.7 | 6.8
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 7.2 | 3.7 | 6 | 2.9 | 2.6 | 6.5
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 1.9 | 3.8 | 1.2 | 3.3 | 8.3 | 11.5
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 12.8 | 11.4 | 6.2 | 4.2 |  | 8.9

24. Secondary Outcome: FSH - Week 24
Description: Lab Values for follicle stimulating hormone
Time Frame: Week 24
Population: FSH measured at Week 24 Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm Data was not collected for patient 24 in placebo-anastrazole-clomiphene arm
Measure: Number; unit: IU/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
IU/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 4.1 | 4.8 | 3 | 5.2 | 6.5 | 4
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 4.4 | 15.1 | 6 | 3.7 | 5.2 | 14.5
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 2 | 7.2 |  | 7.2 | 5.9 | 10.4
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 4.8 | 29.7 | 5 | 5.8 |  |

25. Secondary Outcome: Free Testosterone - Screen
Description: Measure of Free Testosterone
Time Frame: Baseline
Population: FT measured at initial encounter
  Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 18 in placebo-anastrazole-clomiphene arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 8.4 | 6.99 | 7.28 | 8.82 | 6.27 | 7.86
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 6.74 | 9.31 | 6.07 | 9.9 | 5.82 | 5.78
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0
  Patients 13-18 | 9.56 | 12.27 |  | 4.86 | 9.49 |
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 2.19 | 7.27 | 6.52 | 7.71 |  | 6.33

26. Secondary Outcome: Free Testosterone - Week 8
Description: Measure of Free Testosterone
Time Frame: Week 8
Population: FT measured at the end of Week 8 Data was not collected for patient 8 in anastrazole-placebo-clomiphene arm Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 18 in placebo-anastrazole-clomiphene arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 3 | 3
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 19.46 | 21.8 | 17.72 | 35.27 | 2.71 | 12.3
  Patients 7-12: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1
  Patients 7-12 | 15.63 |  | 19.33 | 27.79 | 9.4 | 5.3
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0
  Patients 13-18 | 21.61 | 15.18 |  | 21.71 | 8.91 |
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 17.44 | 20.01 | 11.37 | 15.71 |  | 6.04

27. Secondary Outcome: Free Testosterone - Week 16
Description: Measure of Free Testosterone
Time Frame: Week 16
Population: FT measured at the end of Week 16
  Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 22 in clomiphene-placebo-anastrazole arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 3 | 4
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 14.16 | 16.37 | 12.27 | 12.67 | 19.21 | 17.47
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 8.83 | 5.7 | 14.7 | 9.63 | 14.57 | 13.47
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 10.17 | 5.98 |  | 6.63 | 16.38 | 7.58
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 1
  Patients 19-24 | 14.98 | 9.46 | 11.22 |  |  | 11.62

28. Secondary Outcome: Free Testosterone - Week 24
Description: Measure of Free Testosterone
Time Frame: Week 24
Population: FT measured at the end of Week 24 Data not collected for patient 8 in APC arm Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 18 in placebo-anastrazole-clomiphene arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm No data collected pt 24 in PAC arm
Measure: Number; unit: ng/dl
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 3 | 2
ng/dl
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 10.51 | 19.35 | 6.25 | 11.28 | 8.65 | 19.31
  Patients 7-12: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1
  Patients 7-12 | 6.11 |  | 11.09 | 17.89 | 11.63 | 25.27
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0
  Patients 13-18 | 11.82 | 13.74 |  | 18.19 | 15.49 |
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 5.82 | 13.54 | 6.11 | 16.82 |  |

29. Secondary Outcome: Estradiol - Screen
Description: Measurement of Estradiol levels at initial encounter and at the end of Weeks 8, 16, and 24
Time Frame: Baseline
Population: Estradiol measurement at initial encounter
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: pg/mL
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
pg/mL
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 21.6 | 8.1 | 9.6 | 13.5 | 15.9 | 18.4
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 9 | 19.3 | 21.3 | 11.4 | 18.6 | 10.9
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 13.3 | 20.1 | 16.2 | 14.1 | 15.9 | 13.1
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 9.5 | 15.5 | 26.6 | 11 |  | 26.8

30. Secondary Outcome: Estradiol - Week 8
Description: Measurement of Estradiol levels at initial encounter and at the end of Weeks 8, 16, and 24 An entered value of 4.9 means the measure was <5
Time Frame: Week 8
Population: Estradiol measurement at the end of Week 8
  Data was not collected for patient 2 in anastrazole-placebo-clomiphene arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: pg/mL
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4
pg/mL
  Patients 1-6: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1
  Patients 1-6 | 11.2 |  | 49.8 | 94.5 | 20.8 | 22.5
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 7 | 15.1 | 70.1 | 45 | 18.5 | 9.3
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 9.7 | 4.9 | 25.1 | 33.5 | 10 | 15.9
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 7.4 | 10.7 | 51.7 | 39.1 |  | 27.4

31. Secondary Outcome: Estradiol - Week 16
Description: as for outcome 30
Time Frame: Week 16
Population: Estradiol measurement at the end of Week 16 Data was not collected for patient 2 in anastrazole-placebo-clomiphene arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: pg/mL
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4
pg/mL
  Patients 1-6: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1
  Patients 1-6 | 39.5 |  | 8.9 | 17.9 | 56.9 | 5
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 13.1 | 21.6 | 12.8 | 14.4 | 28.2 | 6.8
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 20.1 | 15 | 23.8 | 13.1 | 37 | 4.9
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 48.5 | 28.3 | 14.8 | 15.9 |  | 4.9

32. Secondary Outcome: Estradiol - Week 24
Description: as for outcome 30
Time Frame: Week 24
Population: Estradiol measurement at the end of Week 24
  Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm Data was not collected for patient 24 in placebo-anastrazole-clomiphene arm
Measure: Number; unit: pg/mL
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
pg/mL
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 22.5 | 43.9 | 16.2 | 9.5 | 18.1 | 41.1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 12.5 | 49.1 | 6.6 | 5 | 11.6 | 85.9
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 25.5 | 36.4 |  | 9.2 | 4.9 | 29.3
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 22.2 | 39.4 | 19 | 4.9 |  |

33. Secondary Outcome: SHBG - Screen
Description: Lab Measure of sex hormone binding globulin at the initial encounter and at the ends of week 8, 16, and 24
Time Frame: Baseline
Population: SHBG measured at initial encounter
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: nmol/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
nmol/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 13.9 | 35.2 | 20 | 31.7 | 26.2 | 24.1
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 30.7 | 12.6 | 23.5 | 26.4 | 20.9 | 26.8
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 23.5 | 17.5 | 21.4 | 20 | 16.9 | 14.8
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 28.6 | 22 | 35.5 | 11.6 |  | 30.6

34. Secondary Outcome: SHBG - Week 8
Description: Lab Measure of sex hormone binding globulin at the initial encounter and at the ends of week 8, 16, and 24
Time Frame: Week 8
Population: SHBG measured at week 8
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: nmol/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
nmol/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 10 | 38.2 | 18.4 | 29.8 | 23.9 | 21.6
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 23.4 | 12.7 | 26 | 27.2 | 24.1 | 25.7
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 26.9 | 16.1 | 21.6 | 30.9 | 14.3 | 17.6
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 28.1 | 20.1 | 42.7 | 20.9 |  | 30.7

35. Secondary Outcome: SHBG - Week 16
Description: Lab Measure of sex hormone binding globulin at the initial encounter and at the ends of week 8, 16, and 24
Time Frame: Week 16
Population: SHBG measured at week 16
  Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm
Measure: Number; unit: nmol/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
nmol/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 22.3 | 35.5 | 13.8 | 16.4 | 33.3 | 17.7
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 30.7 | 15.3 | 26.6 | 31 | 16.7 | 23
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 13-18 | 26.8 | 17.2 | 14.2 | 22.8 | 17.2 | 16.6
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 39.3 | 24.8 | 35 | 13.9 |  | 31

36. Secondary Outcome: SHBG - Week 24
Description: Lab Measure of sex hormone binding globulin at the initial encounter and at the ends of week 8, 16, and 24
Time Frame: Week 24
Population: SHBG measured at week 24
  Data was not collected for patient 15 in clomiphene-anastrazole-placebo arm Data was not collected for patient 23 in placebo-clomiphene-anastrazole arm Data was not collected for patient 24 in placebo-anastrazole-clomiphene arm
Measure: Number; unit: nmol/L
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3
nmol/L
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 14.6 | 41.8 | 15.1 | 25.2 | 29.7 | 23.6
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 7-12 | 33.8 | 16 | 24.4 | 25.3 | 13.8 | 34.1
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 29 | 21.7 |  | 20.1 | 17.3 | 17.5
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0
  Patients 19-24 | 23.2 | 26 | 33.8 | 13.7 |  |

37. Secondary Outcome: SEP #1-3 Cumulative - Screen
Description: Questions 1, 2, and 3 for the Sexual Encounter Profile have been cumulatively added. 1 - yes and 0 - no have been added for questions 1-3 to determine a total value from 0-3.
  0-3: cumulative score from SEP questions 1, 2, and 3
  Higher values (3) are considered to be a better outcomes relative to lower numbers (0) 3 is better than 2 is better than 1 is better than 0
Time Frame: Baseline
Population: SEP measured at the initial encounter
  Baseline SPEP was not measured for participants 1-24
  Table included for completeness
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: SEP #1-3 Cumulative - Week 8
Description: as for outcome 37
Time Frame: Week 8
Population: SEP measured at the end of week 8
  data not collected for pt 11,17 in PCA arm data not collected for pt 13 in ACP arm data not collected for pt 15 in CAP arm data not collected for pt 22 in CPA arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 2 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Patients 1-6 | 3 | 3 | 1 | 1 | 3 | 4
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 7-12 | 2 | 3 | 2 | 2 |  | 3
  Patients 13-18: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 1
  Patients 13-18 |  | 2 |  | 1 |  | 2
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 1
  Patients 19-24 | 3 | 3 | 3 |  | 1 | 2

39. Secondary Outcome: SEP #1-3 Cumulative - Week 16
Description: as for outcome 37
Time Frame: Week 16
Population: SEP measured at the end of week 16
  data not collected for pt 3,15 in CAP arm data not collected for pt 5,11,23 in PCA arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 1 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1
  Patients 1-6 | 2 | 3 |  | 1 |  | 2
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 7-12 | 3 | 3 | 3 | 3 |  | 0
  Patients 13-18: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 | 4 | 3 |  | 3 | 3 | 2
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 19-24 | 3 | 3 | 3 | 3 |  | 1

40. Secondary Outcome: SEP #1-3 Cumulative - Week 24
Description: as for outcome 37
Time Frame: Week 24
Population: SEP measured at the end of week 24 data not collected for pt 1,13 in ACP arm data not collected for pt 3, 15 in CAP arm data not collected for pt 22 in CPA arm data not collected for pt 11,23 PCA arm
Measure: Number; unit: score on a scale
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
Number analyzed (Participants) | 2 | 4 | 2 | 3 | 2 | 4
score on a scale
  Patients 1-6: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 1
  Patients 1-6 |  | 3 |  | 3 | 3 | 2
  Patients 7-12: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1
  Patients 7-12 | 3 | 3 | 3 | 1 |  | 0
  Patients 13-18: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 1
  Patients 13-18 |  | 3 |  | 2 | 0 | 2
  Patients 19-24: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 1
  Patients 19-24 | 3 | 3 | 3 |  |  | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the first dose of medication and at the end of week 8, week 16, and week 24 at a participant and provider meeting.
Description: The 6 arms are comprised of certain orders of drug administration. To maintain the integrity of this order, AE have been listed as part of the arm it belongs to. Details regarding when the AE occurred in relation to the drug being administered at that point in time during the arm is listed at the bottom of the table.
Arm/Group | Anastrazole-clomiphene-placebo | Anastrazole-placebo-clomiphene | Clomiphene-anastrazole-placebo | Clomiphene-placebo-anastrazole | Placebo-clomiphene-anastrazole | Placebo-anastrazole-clomiphene
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 1/4 | 1/4 | 1/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrazole-clomiphene-placebo (N=4) | Anastrazole-placebo-clomiphene (N=4) | Clomiphene-anastrazole-placebo (N=4) | Clomiphene-placebo-anastrazole (N=4) | Placebo-clomiphene-anastrazole (N=4) | Placebo-anastrazole-clomiphene (N=4)
Lyme Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — AE occured during placebo
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrazole-clomiphene-placebo (N=4) | Anastrazole-placebo-clomiphene (N=4) | Clomiphene-anastrazole-placebo (N=4) | Clomiphene-placebo-anastrazole (N=4) | Placebo-clomiphene-anastrazole (N=4) | Placebo-anastrazole-clomiphene (N=4)
Headache (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 — AE occured during anastrazole in both trial arms indicated.
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Osteopenia AE occurred during anastrazole.
Rib Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 — AE occured during anastrazole.
Nasal Septal Deviation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Nasal Septal deviation AE occured during clomiphene.
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Left shoulder AE occured during placebo.
Upper Respiratory Infection (URI) (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 — AE occured during placebo.
Vitamin D deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 — AE occured during placebo.
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — AE occured during clomiphene
Insomnia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 — AE occured during anastrazole in the trial arms indicated.
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 — AE occured during clomiphene of both trial arms indicated
Weight Gain (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 — AE occured during anastrazole
Decreased Libido (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 — AE occured during clomiphene
Bloated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — AE occured during clomiphene
Chronic Maxillary Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — AE occured during clomiphene
Right Big Toe Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 — AE occured during anastrazole
Ringworm (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — Ringworm AE occured during clomiphene.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03933618/Prot_SAP_000.pdf